



Learning from Heart Failure Nurses and Patients: Exploring their Perspectives in the management of depression and anxiety in primary care settings

**Protocol Date: 20.08. 2020** 

Introduction

Heart failure (HF) is a complex clinical syndrome manifested by serious and progressive signs

and symptoms. It is characterized by inability of the heart muscle to pump enough blood to

meet body's blood and oxygen requirements (American Heart Association, 2017). According

to the European Society of Cardiology (ESC) (ESC, 2016) heart failure (HF) is a clinical

syndrome that results in decreased cardiac output and may be accompanied with high

intracardiac pressure during rest or with stress (ESC, 2016). HF induces many changes in a

person's life affecting activities of daily living including breathlessness, chest pain and fatigue

with limited exercise tolerance affecting their ability to function independently.

With increased life expectancy and an aging population, the prevalence of HF is increasing

worldwide. The estimated number of the prevalence of HF cases from 2002 to 2014, increased

by 23% in United Kingdom (UK) (Conrad, 2018). As per the hospital diagnoses, estimates

show that there are up to 920,000 people living with HF in the UK (British Heart Foundation,

2018). In year 2017-2018 in England, 500,000 people were diagnosed with heart failure (NHS

Digital, 2018). Moreover, the ESC published that the prevalence of HF in developed countries

is around 1-2 % among adults and is rising up (≥10%) among people over 70 years of age. It

also indicated that at the age of 55 years, the lifetime risk of developing HF is 33% for males

and 28% for females (ESC, 2016).

With the increased prevalence of HF, there is increased cost of HF related healthcare services,

as HF hospitalization place a major burden on healthcare services worldwide. The overall

management of HF and the frequency of hospital admission leads to increased healthcare

expenditure and cost (Farre, 2016; & Lesyuk, 2018). AHA predicted that with the ageing

population, this disease may reach epidemic proportions (American Heart Association, 2017).

This will increase the healthcare burden as the cost of proving quality care to HF patients is

ranked among the leading healthcare expenditures in the US (American Heart Association,

2017). In United Kingdom, the increased utilization of medical services places an extra burden

on the NHS budget as it costs more than £2 billion a year (BHF, 2016).

The physiological symptoms of HF such as breathlessness can lead to increased hospitalization.

Due to the pathological changes induced in HF, many patients develop depression and anxiety.

Anxiety is unpleasant feelings of unease, worry or fear that many people experience, and cause negative emotions and thinking (Tully *et al.*, 2014). Anxiety is a normal feeling unless it becomes constant or when anxious people fail to control their worries and it starts affecting their daily lives (Wells, 2018b). Symptoms of anxiety can be physical and include restlessness, sleeping difficulties and palpitations (Palacios *et al.*, 2018). For those with HF, they may become anxious due to the activity limiting symptoms of their HF and the associated breathlessness. Anxiety disorder were found to be responsible for adverse outcomes in coronary artery disease but the association between it and HF is less clear (Celona, 2018) and was under-researched. Therefore, in this study anxiety will be explored in HF.

Depression is a common comorbidity in HF due to the pathological similarities between both conditions. With depression, patients are unable to carry out activities of daily living or to function at home or work for at least two weeks (Lesperance & Frasure-Smith, 2000). Depression is considered as a treatable serious medical illness that negatively affects the way people feel, think or even they act, and it can be classified as mild, moderate or severe. Depression may lead to loss of interest in activities, appetite change, changes in sleep pattern, increased fatigue, feeling worthless and hopeless, difficulty in concentration and developing ideas of attempting suicide (Halaris, 2009; Frasure-Smith & Lesperance, 2010). Many HF patients develop depression and the prevalence of depression found to steadily increase from 11% to 42% as the class of New York Heart Association (NYHA) functional status increases from I to IV (Silver, 2010) (i.e. patients become more symptomatic with HF and their prognosis worsens).

The American Heart Association (AHA) (ACCF & AHA, 2013) guidelines on depression and coronary heart disease recommended the consideration of depression as an independent risk factor for poor prognosis in acute coronary syndrome which is known as a leading cause of HF (Lichtman et al, 2014). Also, the AHA HF guidelines considered depression as a common and important comorbidity in HF that can lead to poorer clinical outcomes and poor Health-Related Quality of Life (HRQOL) (ACCF & AHA, 2013).

Studies (Marti, 2013; Sherwood, 2011; Nieminen, 2015; Gheorghiade, 2013; Moraska, 2013; Wallenborn, 2013; & Hawkins, 2013) have reported that depression is associated with increased hospitalization and death and worsens clinical outcomes in HF. Depression in HF also found to be closely associated with increased outpatients and emergency department visits

Version 2.1, Date: 20.8.2020


(Moraska, 2013) and of all-cause mortality (Gathright, 2017; Moraska, 2013; Freedland, 2016;

& Adelborg, 2016). Moreover, patients with worsening depressive symptoms were found to be

at higher risk of death for up to one year following hospital discharge (Freedland, 2016).

Studies (Gottlieb, 2004; & Hwang, 2014) also reported that Quality of Life (QOL) scores were

significantly worse for HF patients with depression. The evidence clearly showed that

depression in HF increases healthcare expenditure and cost (Wallenborn, 2013). Therefore, it

is crucial to effectively detect and manage depression in HF that may lead to improvement in

QOL and improved life expectancy.

The ESC HF guidelines highlighted the importance of routine depression screening with a

validated questionnaire. It also emphasized on initiating treatment for depression for all heart

failure patients including the use of psychosocial interventions, pharmacological therapy or

exercise training (ESC, 2016).

The National Institute for Health and Care Excellence (NICE) guidelines (NICE, 2016) on

heart failure emphasized the importance of treating depression in heart failure but there were

no specific treatment options for HF recommended in the document (NICE, 2016). Due to the

clinical effects of depression in HF, it is important to effectively assess and treat depression as

remission from depression found to improve outcomes (Jiang, 2011). In Southwark and

Lambeth, inpatients diagnosed with HF are being assessed for depression. The community-

based HF patients are being assessed for anxiety and depression using PHQ-9 and GAD-7.

However, the frequency and the process of assessment need to be further explored. The HF

community nurses works through the KHP partnership with Guy's and St. Thomas's and King's

College Hospital to provide the integrated heart failure service in the local area of Southwark

and Lambeth in South London. The integrated heart failure team consists of heart failure

specialist community nurses and consultant cardiologist with two pharmacists (Guy's and St

Thomas' NHS Foundation Trust, 2019). The service provides specialist care in both the hospital

and community with support for GPs on HF diagnosis and management. The aim of the

integrated heart failure team in the community is to provide the HF treatment effectively, help

patients understand and manage their symptoms and support with lifestyle changes.

Even though, the community HF nurses have extensive role in managing HF patients in the

community, their role in assessing anxiety and depression; and providing psychological

treatment need to be further explored. The community-based HF patients who are diagnosed with depression are usually referred for psychological treatment (IAPT or 3DLC). The type of treatment depends on the severity of their depression and the extent to which depression is affecting clients' self-management of HF. So, for persistent and mild to moderate depression or if the depression is not related to HF, the patients will be referred for Improving Access for Psychological Therapies (IAPT) for treatment. While, for moderately severe to severe depression and whose depression affects their management of HF, patients will be seen by the team of 3 Dimensions for Long Term Conditions (3DLC). However, the process of providing treatment and type of therapy offered is not known and need to be further explored.

The London Cardiac Clinical Network (LCCN) in 2017 recommended that all HF services (in hospital and the community) must be knowledgeable regarding the process of referring patients to specialist services including IAPT and should understand the local pathway for referral. Based on this, they recommended that Commissioners must ensure the availability of community services for HF patients that can optimize the medical therapy, provide self- care support, psychosocial support and exercise-based rehabilitation. The LCCN also recommended that secondary care heart failure specialist should have direct access to these services. Support from the LCCN in 2017/18 and 2018/19 reported that follow-up and community care can be improved by enhancing collaboration with the London Mental Health Clinical Network in order to upskill healthcare professionals in IAPT services thus can support people with HF and depression. Also, by promoting an understanding to those working in HF services of local pathways for referral to specialist IAPT services. (LCCN, 2017). This will enable the community HF nurses to be able to provide holistic care which includes physical, mental and social care needs.

Unfortunately, the current literature shows the gap in depression and anxiety assessment and treatment in the community. Therefore, there is a need to assess the process by which community HF nurses assess and manage depression and anxiety. This current study builds on our recent systematic review (phase 1) (Helal, *et al*, submitted) which illustrated that CBT could be effective in improving depressive symptoms in HF, but more studies are needed to build on these findings. The findings from this review will be used in this current study to examine how community HF nurses are assessing, managing and treating depression and anxiety in community-based HF patients. Also, to identify community-based HF patients' views and experiences regarding depression and anxiety assessment and treatment.


Study objectives and purpose

In this current study, online focus group and qualitative telephone/online interviews will be

undertaken to explore the community heart failure nurses' and community-based HF patients'

views and experiences in managing depression and anxiety; and to assess whether COMPASS

a web-based intervention would be useful.

With the COVID-19 pandemic extra measures were taken to protect HF patients who are

considered as clinically vulnerable (shielding). This impacted on patients access to treatment

and health care services, community networks and support from family and friends. It is

anticipated during the pandemic this has had a deleterious impact on individuals' mental health

with increased social isolation, anxiety about care and treatment, and risk of poor outcome if

contract COVID-19. This study will explore the impact of COVID-19 on the psychological

wellbeing of community-based HF patients.

**Research Question** 

How is depression and anxiety being assessed, managed and treated in community-based HF

patients; and what is their views on the use of web-based intervention?

**6.1. Aims** 

To explore community HF nurses' and patients' views and experiences in managing

depression and anxiety and to assess whether COMPASS a web-based intervention would be

a useful intervention.

**Primary objective** 

To explore community HF nurses' and patients' views and experiences of managing depression

and anxiety and to assess whether COMPASS a web-based intervention would be useful.

Secondary objectives

1) To conduct online focus groups with community HF nurses (n=5) and qualitative

telephone/online interviews with community-based HF patients (n=8) within Lambeth

and Southwark NHS Trusts.

2) To synthesise the data obtained from online focus groups and qualitative telephone/online

interviews using thematic analysis.

3) To understand how depression and anxiety is managed in HF patients and whether web-

based intervention would be a useful intervention.

To explore the impact of COVID-19 on community-based HF patients' depression and anxiety

level changes to management processes.

Study design

A qualitative methodology will be employed using online focus group and qualitative

telephone/online interviews. In this current study online focus group will be undertaken with

community HF nurses (n=5) and qualitative telephone/online interviews with community-

based HF patients (n=8). Online focus group allows for expression of personal opinions,

perspectives and experiences regrading an issue of interest. The synergy of the online focus

group allows participants to collectively brainstorm together, add on others' ideas and this may

provide rich and large amount of opinions, issues and concepts (Brinkmann, 2015).

Even though qualitative telephone interviews are used less frequently than the traditional face-

to-face interviews (Opdenakker, 2006; Sweet, 2002), it can be a useful data collection method

(Carr & Worth, 2001, p. 521). The participants of qualitative telephone interviews were found

to feel more comfortable being interviewed over the telephone and talking more freely than

face to face interviews (Novick, 2008). The qualitative data obtained from telephone interviews

were reported to be rich, comprehensive and of high quality (Chapple, 1999; Kavanaugh &

Ayres, 1998; Sturges & Hanrahan, 2004; Sweet, 2002). In comparison to face-to-face

interviews, the qualitative telephone interviews were less costly (Chapple, 1999), can increase

access to different geographically located participants (Sturges & Hanrahan, 2004; Sweet,

2002; Tausig & Freeman, 1988) and is safer for the interviewer (Carr & Worth, 2001; Sturges

& Hanrahan, 2004). Qualitative telephone interview also allows more anonymity (Sweet, 2002;

Tausig & Freeman, 1988), privacy (Sturges & Hanrahan, 2004), and decrease in social pressure

(McCoyd & Kerson, 2006).

Qualitative methodology was deemed the best method to meet the study aims and to understand

how community HF nurses are assessing, managing and treating depression and anxiety in

community-based HF patients; and what they think of using a web-based Intervention (i.e.

COMPASS). Qualitative methods are a useful method to explore the depth of participants'

views and opinions related to an issue of interest, and to capture participants' interpretations

regarding a concept. Online focus group is useful for the researcher to grasp how those who

take part perceive the process and feel comfortable including experiences and emotions around

a particular topic (Barbour, 2005). Barbour (2005) highlights how focus group enables the

researcher to observe record and analyse the group's interactions to include this in the

presentation of findings.

Subject inclusion criteria

Inclusion criteria for Community-based HF patients:

1) Community-based HF patients with clinically established HF diagnosis (confirmed HF

diagnosis) in Lambeth and Southwark Boroughs who have mild to moderate symptoms

of depression with/without anxiety confirmed by PHQ-9 (5-14) and GAD-7;

2) Patients with NYHA class I-III;

3) Capacity to provide informed consent; and

4) Proficiency in English language so can fully respond to verbal and written material.

Inclusion criteria for Community HF nurses:

1) All community-based HF-nurses employed in Lambeth and Southwark Boroughs who

are registered with Nursing Midwifery Council (NMC) will be invited to participate in

the study;

2) Capacity to provide informed consent;

3) Community HF-nurses who are actively providing care to community-based HF

patients; and

4) have access to internet connected computer or device and technology for Microsoft

(MS) Teams.

Subject exclusion criteria

8.2.1. Exclusion criteria for community-based HF patients:

1. Community-based HF patients under 18 years of age;

2. Participants who are deemed not to have the capacity to consent;

3. Patients with cognitive impairment or dementia confirmed by medical records; and

4. Community-based HF patients with NYHA class IV.

5. Patients with severe depression and/or having suicidal ideation.

Exclusion criteria for Community HF nurses:

1. Nurses working with inpatients or in the OPD departments; and

2. Nurses who are not employed as community HF nurses.

3. Any community HF nurse who do not have access to internet or online technology.

**Study procedures** 

Subject recruitment

A purposive sampling will be used to capture data from community heart failure nurses and

community-based HF patients who meet the inclusion criteria. Participants will be recruited

directly by GSTT community HF services in Southwark and Lambeth Boroughs as they have

an established community HF service.

**Patients recruitment:** 

Participants will be recruited from Guys and St. Thomas's community-based HF services in

Lambeth and Southwark Boroughs through discussion with community HF lead nurse. The

invitation letter and participants information sheets will be sent by email to HF lead nurse and

community HF nurses and they will be asked to identify community-based HF patients to

participate in the study. The information sheets include contact details inviting volunteers to

email or phone the researcher. Alternatively, community-based HF patients who are willing to

participate can give their contact details to the nurses who will send it over to the researcher.

Once this contact is received the researcher will contact possible participants via participant's

preferred method (phone, online or email) to offer the opportunity to discuss what would be

involved in more details and answer any question. Inclusion criteria (described earlier) will be

used to assess eligibility to the study. In addition, the researcher will arrange a time to call back

the participants who are not ready to decide regarding participation in the study.

**Nurse recruitment:** 

The community HF lead nurse will be approached by the researcher via telephone/email to

allow approaching the community HF nurses. Invitation letter and participant information

sheets will be provided by the researcher via email. Participants will be given time to read the

information and respond via email or telephone at which further information on the study will

be provided and any questions will be answered.

Procedure for online focus groups:

The online focus groups with community HF nurses who consent and meet the eligibility for

this study will be conducted by the researcher. The online focus group may take 60-90 minutes

with breaks in between as this time period reported with less participants fatigue (McCoyd and Kerson, 2006). The emphasis will be open-ended form of conversation that can provide opportunities for rich discussions and sharing of personal experiences and interpretations.

The date of the online focus group will be decided according to community HF nurses' preferences. A time will be agreed with their manager when all of the community HF nurses can meet as a group. The PIS and consent form will be sent to all community HF nurses by email. The consent form will be signed ahead of time and gathered online. Similarly, baseline demographic data will be sent and collected online. The community HF nurses will be involved in the online focus group that will be conducted using Microsoft teams. A link to the online focus group will be sent by the researcher to all community HF nurses with the agreed date and time. The online focus group will have a skilled moderator who is the researcher's supervisor

(co-investigator). The moderator will moderate the session and will deal with any arising

technical issues.

The discussion with community HF nurses will include their perspectives about depression and anxiety assessment and management process and what they think of web-based intervention. Then, the community HF nurses will have a short break. Immediately after the break, a COMPASS team member will join the online focus group and will demonstrate the COMPASS web-based intervention to the community HF nurses. Community HF nurses will be allowed to ask questions regarding COMPASS before the COMPASS team member leaves the online focus group. Once demonstration is complete and the COMPASS personnel has left the online focus group, the researcher will take over and will assess community HF nurses' perspectives regarding COMPASS. The participants will be asked if a similar intervention will be useful to community-based HF patients and which aspects of COMPASS they feel is relevant and important in HF. Issues around potential barriers and facilitators for implementation will also

be explored.

Procedure for the Qualitative telephone/online interviews

For the community-based HF patients, qualitative telephone/online interviews will be conducted with each participant at their preferred time and method. Due to COVID-19, the participants will be interviewed in their own home at a time that suits them. Qualitative telephone/online interviews may take 60-90 minutes. The consent form will be sent online to community-based HF patients who have access to the internet and email. Participants who do


not have internet access a recorded consent over the telephone will be obtained. This will be done by the researcher who will read the consent form to the participants and they will be asked for their verbal consent on each statement and their answer will be recorded e.g. Do you agree to...? YES, NO. Once consent is obtained, the researcher will email the community-based HF patients a video link to COMPASS before they engage with qualitative telephone/online interviews. This video link is a demonstration of the COMPASS web-based intervention and the researcher will encourage them to view the video so they can share their views about COMPASS during the qualitative telephone/online interview. For participants who do not have access to email or the internet, the COMPASS will be explained to them by the researcher. They will be encouraged to explore the concept of web-based intervention, what services and resources the clinicians need to consider when introducing web-based interventions to people who do not have access to the internet etc.

At the start of the qualitative telephone/online interviews, rapport will be established with the participant in person (Burke & Miller, 2001; Carr & Worth, 2001) and predeveloped interview script will be used to introduce the study at the beginning of the interview (Burke & Miller, 2001). The discussion with community-based HF patients will include their perspectives about depression and anxiety assessment and management process and what they think of web-based intervention. Then, the participants will be asked about using web-based intervention for the management of depression and anxiety in general and about COMPASS intervention in specific if they have viewed the video. The participants will be asked if they think that a web-based intervention will be applicable to them and if they feel that it can be useful in HF. Also, the community-based HF patients will be asked to identify the potential barriers and facilitators for implementation of any web-based intervention.

## Data to be collected

The demographic form will be sent to community HF nurses and they will be asked to complete and return this via email to the researcher before the online focus group.

The demographic form will also be emailed to community-based HF patients and they will also be asked to complete and return this via email to the researcher before the qualitative telephone/online interview. For community-based HF patients who do not have email access, the researcher will read the information required from the baseline demographic form and will ask them to provide an answer before the interview starts.


Data handling and record keeping

Data collection will include note taking, digital encrypted Dictaphone and remarking

participants' nonverbal cues when possible. The online focus groups using encrypted Microsoft

(MS) teams with community HF nurses will be audio recorded using digital encrypted

Dictaphone. The qualitative telephone/online interviews with community-based HF patients

will be in a private room and will be audio-recorded using digital encrypted Dictaphone. The

participants will be assured that privacy and confidentiality will be maintained, as the

researcher will be sitting alone in a private room during the interview.

Field notes on the group interactions and processes will also be transcribed by the researcher.

Thematic analysis assisted by N-vivo 12 will be used to allow the development and 'saturation'

of themes and categories.

An online consent form will be sent to community HF nurses which will be signed prior to the

scheduled online focus group. For community-based HF patients, the consent form will be

recorded at the start of the interview, and the participant will be asked whether they agree with

each statement read by the researcher e.g. Do you agree to...? YES, NO.

All the online collected consent forms, participants personal data and qualitative data

recordings and transcripts will be encrypted before they are uploaded to a secure and encrypted

cloud storage area provided by KCL and will only be accessible by researcher and the two co-

investigators. Once the study has been completed, the recordings will be destroyed by deleting

them from the encrypted and password protected file sharing cloud.

Sample size:

This study will include five Community HF nurses and eight community-based HF patients,

13 in total (n=13). A total of five community HF nurses (n=5) will be recruited for the online

focus group and eight community-based HF patients (n=8) will be recruited for the qualitative

telephone/online interviews. Online focus group can vary in size but tend to average between

6 to 8 but it is recommended to reduce the number to 4-5 participants for online focus group.

Smaller group size (around six) are advised where the topic is controversial, where the

participants have considerable knowledge or are likely to have strong views on the subject. The

qualitative telephone interviews will include eight community-based HF patients.

**DATA ANALYSIS:** 

The qualitative date from online focus group will be entered into a computer-assisted

qualitative data analysis package (NVivo 12). The verbatim transcription will be conducted for

the audio data obtained from online focus group. Coding will be based on the research

questions as well as emerging themes. Field notes on the online group interactions and

processes will also be transcribed. The qualitative data from qualitative telephone interviews

will be transcribed using NVivo 12. Data Coding will be done, and emerging themes will be

identified.

Thematic analysis will be used to analyse the themes. Final categories and themes will be

determined using a consensus approach to resolve any differences in interpretation. The data

will be managed using NVivo 12 to organise the ongoing analysis, themes and categories.

**Ethical considerations** 

An application to NHS R&D and IRAS is currently under preparation for submission. The

community HF nurses will email the consent form to the researcher before the online focus

group takes place. The community-based HF patients will send the consent form either via

email if they have internet access or they will be consented verbally and recorded at the

beginning of the qualitative telephone/online interview.

During recruitment of the participants, the researcher will discuss the purpose of the study and

the criteria for participation. The researcher will assure all the participants that anonymity will

be provided, and they can withdraw at any time. Participants will also be informed that no harm

will result from taking part in the study or even by refusing to participate. It is not anticipated

that participation in the study will be stressful. However, before the online focus group or

qualitative telephone/online interviews commences, it will be explained to all participants that

they do not have to answer any questions they do not wish to or that make them uncomfortable.

In addition, the online focus group will be co-facilitated by the co-investigator who is a mental

health lecturer with extensive experience in clinical mental health practice and psychological

therapy.

Moreover, it will be clearly explained to all participants that all data will be pseudo-anonymised

during transcription and that data will be stored securely under a study number whereas

comments quoted in any reports, results, published papers or feedback will not be linked to any individual.

## Reporting and dissemination

The study will be published in a peer-reviewed scientific journal.


## References

ACCF &AHA. (2013). 2013 ACCF/AHA Guideline for the Management of Heart Failure. Journal of American College of Cardiology, 62 (16, 147-239.

Adelborg, K., Schmidt, M., Sundboll, J., Pedersen, L., Videbech, P., Botker, H. E., Sorensen, H. T. (2016). Mortality Risk Among Heart Failure Patients with Depression: A Nationwide Population-Based Cohort Study. *J Am Heart Assoc*, *5*(9). doi:10.1161/JAHA.116.004137

American Heart Association (2017). Classes of heart failure. Retrieved from https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure on 29 Dec 2018

American Heart Association (2017). What is Heart Failure? Retrieved from https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure on 24 NOV 2018

American Psychiatric Association (2017). Depression. retrieved from https://www.psychiatry.org/patients-families/depression/what-is-depression on 24 NOV 2018

Barbour, R., S. (2005). Making sense of focus groups. Medical Education, 39 (7), 742-750. https://doi.org/10.1111/j.1365-2929.2005.02200.x

Brinkmann, S., Kvale, A. (2015). *Interviews Learning the Craft of Qualitative Research Interviews*. 3<sup>rd</sup> ed. SAGE, California

British Heart Foundation (2018). UK fact sheets. Retrieved 12.12.2018 from https://www.bhf.org.uk/what-we-do/our-research/heart-statistics on 18 December 2018

Celano, C. M., Villegas, A. C., Albanese, A. M., Gaggin, H. K., & Huffman, J. C. (2018). Depression and Anxiety in Heart Failure: A Review. *Harv Rev Psychiatry*, 26(4), 175-184. doi:10.1097/HRP.0000000000000162

Conrad, N; Judge, A, Tran, J et al. (2018). Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals, The Lancet, 2018; 391, 10120


retrieved from http://www.thelancet.com/journals/lancet/article/PIIS0140-6736(17)32520-5/fulltext?elsca1=tlpr

ESC (2016). 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. *Eur Heart J, 37*(27), 2129-2200. doi:10.1093/eurheartj/ehw128

Farre, N., Vela, E., Cleries, M., Bustins, M., Cainzos-Achirica, M., Enjuanes, C., Moliner, P., Ruiz, S., Verdu-Rotellar, J.M. & Comin-Colet, J. (2016) Medical resource use and expenditure in patients with chronic heart failure: a population-based analysis of 88 195 patients. *Eur J Heart Fail*, 18(9), 1132-40.

Frasure-Smith N., Lesperance F. (2010). Depression and cardiac risk: present status and future directions. Heart 96, 173–176. 10.1136/hrt.2009.186957

Freedland, K. E., Hesseler, M. J., Carney, R. M., Steinmeyer, B. C., Skala, J. A., Davila-Roman, V. G., & Rich, M. W. (2016). Major Depression and Long-Term Survival of Patients With Heart Failure. *Psychosom Med*, 78(8), 896-903. doi:10.1097/PSY.

Gathright, E.C., Goldstein, C.M., Josephson, R.A. & Hughes, J.W. (2017) Depression increases the risk of mortality in patients with heart failure: A meta-analysis. *Journal of Psychosomatic Research*, 94, 82-89

Gheorghiade, M., Vaduganathan, M., Fonarow, G. C., & Bonow, R. O. (2013). Rehospitalization for heart failure: problems and perspectives. *J Am Coll Cardiol*, *61*(4), 391-403. doi:10.1016/j.jacc.2012.09.038

Gottlieb, S. S., Khatta, M., Friedmann, E., Einbinder, L., Katzen, S., Baker, B., Thomas, S. A. (2004). The influence of age, gender, and race on the prevalence of depression in heart failure patients. *J Am Coll Cardiol*, *43*(9), 1542-1549. doi:10.1016/j.jacc.2003.10.064


Guy's and St Thomas' NHS Foundation Trust, 2019. Integrated heart failure service (community): Providing heart failure care in Southwark and Lambeth retrieved on 25<sup>th</sup> June 2019 from https://www.guysandstthomas.nhs.uk/our-services/community-heart-failure/overview.aspx

Halaris A. (2009). Comorbidity between depression and cardiovascular disease. Int. Angiol. 28, 92–99.

Hawkins, N. M., Wright, D. J., & Capewell, S. (2013). Heart failure services in the United Kingdom: rethinking the machine bureaucracy. *Int J Cardiol, 162*(3), 143-148. doi:10.1016/j.ijcard.2011.10.144

Helal, S., I., Lee, G., Grealish, A. (submitted). The Efficacy of Psychological interventions on health-related quality of life for chronic heart failure patients with depression: A Systematic Review *(in process)* 

Hwang, S. L., Liao, W. C., & Huang, T. Y. (2014). Predictors of quality of life in patients with heart failure. *Jpn J Nurs Sci*, 11(4), 290-298. doi:10.1111/jjns.12034

Jiang, W., Krishnan, R., Kuchibhatla, M., Cuffe, M.S., Martsberger, C., Arias, R.M., O'Connor, C.M. & Investigators, S.-C. (2011) Characteristics of depression remission and its relation with cardiovascular outcome among patients with chronic heart failure (from the SADHART-CHF Study). *Am J Cardiol*, 107(4), 545-51.

Lesperance F., Frasure-Smith N. (2000). Depression in patients with cardiac disease: a practical review. J. Psychosom. Res. 48, 379–391. 10.1016/S0022-3999(99)00102-6

Lesyuk, W., Kriza, C. & Kolominsky-Rabas, P. (2018) Cost-of-illness studies in heart failure: a systematic review 2004-2016. *BMC Cardiovasc Disord*, 18(1), 74.

Lichtman, J.H., Froelicher, E.S., Blumenthal, J.A., Carney, R.M., Doering, L.V., Frasure Smith, N., et al. (2014). Depression as a risk factor for poor prognosis among patients with acute coronary syndrome: systematic review and recommendations: a scientific statement from the American Heart Association. Circulation 129 (12),1350–1369


London Cardiac Clinical Network (2017). Improving heart failure services for people in London Review, recommendations and offer of support from the London Cardiac Clinical Network. Retrieved on 25<sup>th</sup> June 2019 from http://www.londonscn.nhs.uk/wp-content/uploads/2017/07/Improving-heart-failure-services-for-people-in-London.pdf Marti, C.N., Fonarow, G.C., Gheorghiade, M. & Butler, J. (2013) Timing and duration of interventions in clinical trials for patients with hospitalized heart failure. *Circ Heart Fail*, 6(5), 1095-101.

Moraska, A. R., Chamberlain, A. M., Shah, N. D., Vickers, K. S., Rummans, T. A., Dunlay, S. M., . . . Roger, V. L. (2013). Depression, healthcare utilization, and death in heart failure: a community study. *Circ Heart Fail*, *6*(3), 387-394. doi:10.1161/CIRCHEARTFAILURE.112.000118

NHS Digital (2018). Quality & Outcomes Framework prevalence data. Retrieved 12.12.2018 from https://digital.nhs.uk/data-and-information/publications/statistical/quality-and-outcomes-framework-achievement-prevalence-and-exceptions-data

NICE (2016). Chronic heart failure in adults: management. Retrieved from https://www.nice.org.uk/guidance/cg108 on 11 October 2018

NICE (2016). Depression in adults with a chronic physical health problem: recognition and management. Retrieved from https://www.nice.org.uk/guidance/cg91 on 11 October 2018

NICE (2016). Depression in adults: recognition and management. Retrieved from https://www.nice.org.uk/guidance/cg90/resources/depression-in-adultsrecognition and-management-975742636741 on 11 October 2018

Nieminen, M. S., Dickstein, K., Fonseca, C., Serrano, J. M., Parissis, J., Fedele, F., Zymlinski, R. (2015). The patient perspective: Quality of life in advanced heart failure with frequent hospitalisations. *Int J Cardiol, 191*, 256-264. doi:10.1016/j.ijcard.2015.04.235

Palacios J., Khondoker M., Mann A., Tylee A., Hotopf M. (2018). Depression and anxiety symptom trajectories in coronary heart disease: Associations with measures of disability and


impact on 3-year health care costs. J. Psychosom. Res. 104, 1–8. 10.1016/j.jpsychores.2017.10.015

Ritchie, J. & Spencer, L. 1994. Qualitative data analysis for applied policy research by Jane Ritchie and Liz Spencer in A. Bryman and R. G. Burgess [eds.] 'Analysing qualitative data', (pp.173-194). London: Routledge.

Sherwood, A., Blumenthal, J.A., Hinderliter, A.L., Koch, G.G., Adams, K.F., Jr., Dupree, C.S., Bensimhon, D.R., Johnson, K.S., Trivedi, R., Bowers, M., Christenson, R.H. & O'Connor, C.M. (2011) Worsening depressive symptoms are associated with adverse clinical outcomes in patients with heart failure. *J Am Coll Cardiol*, 57(4), 418-23

Silver, M. A. (2010). Depression and heart failure: An overview of what we know and don't know. *Cleveland Clinic Journal of Medicine*, 77 Suppl 3, S7-S11. doi:10.3949/ccjm.77.s3.02

Tully P. J., Cosh S. M., Baumeister H. (2014). The anxious heart in whose mind? A systematic review and meta-regression of factors associated with anxiety disorder diagnosis, treatment and morbidity risk in coronary heart disease. J. Psychosom. Res. 77, 439–448. 10.1016/j.jpsychores.2014.10.001

Wallenborn, J., & Angermann, C. E. (2013). Comorbid depression in heart failure. *Herz*, *38*(6), 587-596. doi:10.1007/s00059-013-3886-

Wallenborn, J., & Angermann, C. E. (2013). Comorbid depression in heart failure. *Herz*, *38*(6), 587-596. doi:10.1007/s00059-013-3886-

Wells A., McNicol K., Reeves D., Salmon P., Davies L., Heagerty A., et al. (2018b). Metacognitive therapy home-based self-help for cardiac rehabilitation patients experiencing anxiety and depressive symptoms: study protocol for a feasibility randomised controlled trial (PATHWAY Home-MCT). Trials 19:444. 10.1186/s13063-018-2826-x

Burke, L.; Miller, M. Phone interviewing as a means of data collection: Lessons learned and practical recommendations [Online journal]. Forum: Qualitative Social Research. 2001.


Retrieved August 28, 2007 from http://www.qualitative-research.net/fqs-texte/2-01/2-01burkemiller-e.htm

Carr EC, Worth A. The use of the telephone interview for research. NT Research. 2001; 6:511–524.

Opdenakker, R. Advantages and disadvantages of four interview techniques in qualitative research [Electronic Journal]; Forum: Qualitative Social Research. 2006. p. Article 11Retrieved August 28, 2007 from http://www.qualitative-research.net/fqs-texte/4-06/06-4-11-e.htm

Novick, G., (2008). Is There a Bias Against Telephone Interviews In Qualitative Research?. Res Nurs Health, 31(4): 391–398. doi:10.1002/nur.20259.

Chapple, A. Nurse Researcher. Vol. 6. 1999. The use of telephone interviewing for qualitative research; p. 85-93. Retrieved from Journals@OVID

Kavanaugh K, Ayres L. "Not as bad as it could have been": Assessing and mitigating harm during research interviews on sensitive topics. Research in Nursing & Health. 1998; 21:91–97. [PubMed: 9472241]

Sturges JE, Hanrahan KJ. Comparing telephone and face-to-face qualitative interviewing: A research note. Qualitative Research. 2004; 4:107–118.

Sweet L. Telephone interviewing: Is it compatible with interpretive phenomenological research? Contemporary Nurse. 2002; 12:58–63. [PubMed: 12013519]

Tausig JE, Freeman EW. The next best thing to being there: Conducting the clinical research interview by telephone. American Journal of Orthopsychiatry. 1988; 58:418–427. [PubMed: 3407732]

McCoyd JL, Kerson TS. Conducting intensive interviews using email: A serendipitous comparative opportunity. Qualitative Social Work. 2006; 5:389–406.

